CLINICAL TRIAL: NCT05712538
Title: A Study in Two Parts: (Phase 1) A Randomized, Double-blinded, Placebo--controlled, Single-ascending-dose Study in Healthy Adult Subjects and (Phase 1b) an Open-label, Nested, Divided-dose Study in Adults With Cystic Fibrosis to Assess the Safety, Tolerability, and Pharmacokinetics of ARCT-032
Brief Title: Safety, Tolerability, and Pharmacokinetics of ARCT-032 in Healthy Adult Subjects and Adults With Cystic Fibrosis.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Arcturus Therapeutics, Inc. (Industry)
Collaborators: Novotech CRO (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ARCT-032-01
Record Dates: First submitted 2023-01-26; First posted 2023-02-03 (Actual); Last update posted 2024-11-13 (Actual); Status verified 2024-11

CONDITIONS: Cystic Fibrosis
Keywords: Cystic Fibrosis, CF
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Intervention Model Description: Double-blind, placebo controlled (Phase 1 only)
Who Masked: Participant, Investigator
Masking Description: Participant and investigator masking only applies to Phase 1 healthy volunteers only. For Phase 1b, there is no masking, None (Open Label) should be applied.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- ARCT-032, Healthy Adults (Experimental): Ascending single doses of ARCT-032 administered to healthy adults via nebulizer
  Interventions: Drug: ARCT-032
- Placebo, Healthy Adults (Placebo Comparator): Single doses of 0.9% Saline administered to healthy adults via nebulizer
  Interventions: Other: Placebo
- ARCT-032,. Adults with Cystic Fibrosis (Experimental): Two doses of ARCT-032 administered to adults with Cystic Fibrosis via nebulizer
  Interventions: Drug: ARCT-032

INTERVENTIONS:
Drug: ARCT-032 — ARCT-032 is messenger RNA (mRNA) coding for cystic fibrosis transmembrane conductance regulator (CFTR) protein, formulated in a lipid nanoparticle (LNP).
  Arms: ARCT-032, Healthy Adults; ARCT-032,. Adults with Cystic Fibrosis
Other: Placebo — Normal saline
  Arms: Placebo, Healthy Adults

SUMMARY:
Determine the safety, tolerability and pharmacokinetics of single doses of ARCT-032 in healthy adult subjects (Phase 1) and of two doses in Adults with Cystic Fibrosis (Phase 1b).

DETAILED DESCRIPTION:
Phase 1 of this study is a single ascending dose, first-in-human study to determine the safety, tolerability, and pharmacokinetics (PK) of ARCT-032. After screening, healthy adult participants will be randomized 3:1 to inhale a single dose of nebulized ARCT-032 or placebo. There are 4 planned sequential dose cohorts. After dosing, participants will have follow-up assessments over a 4-week period.

Phase 1b in adults with cystic fibrosis will enroll after Phase 1 is completed and safety data are reviewed. Phase 1b is an open-label, two-dose study in adults with cystic fibrosis to assess the safety, tolerability, and pharmacokinetics of ARCT-032. After completion of screening, each participants will inhale two doses of nebulized ARCT-032 two days apart. Participants will have follow-up assessments over a 4-week period.

ELIGIBILITY:
Key Inclusion Criteria:

1. Phase 1: Healthy males or females aged 18 to 65 years at the time of informed consent.

   Phase 1b: Males or females aged 18 to 65 years with confirmed diagnosis of CF documented in subject's medical record
2. Body weight between 40-100Kg and body mass index between 16-35 kg/m2
3. Phase 1: Forced expiratory volume (FEV1) at screening >85% of predicted value for age, sex, and height.

   Phase 1b: FEV1 at screening between 50% and 100% of predicted value
4. Surgically sterile or using an acceptable contraceptive method from the time of signing the informed consent form until at least 30 days after the last dose of study drug.
5. Phase 1b only: Subjects with CF on CFTR modulator therapy must be on a stable regimen for at least 2 months prior to screening.

Key Exclusion Criteria:

1. History of illness or condition that might pose an additional risk or may confound study results.
2. Pregnant or lactating (breast feeding)
3. History of severe allergic reaction to a liposomal product
4. Clinically significant abnormalities in Screening laboratory results
5. Known history of or positive test for human immunodeficiency virus (HIV), hepatitis C or chronic hepatitis B
6. Treatment with another investigational drug, biological agent, or device within 30 days of screening, or 5 half-lives of investigational drug, whichever is longer
7. Drug or alcohol abuse within the past year
8. History of moderate to heavy smoking or vaping (>10 cigarettes/sessions per day) within 6 months prior to the dose of study drug. Participants must be willing to refrain from smoking or vaping within 1 week of dosing through Day 15
9. Systemic or inhaled corticosteroids within 3 months prior to screening (Phase 1 only).
10. Have any other conditions, which, in the opinion of the Investigator or Sponsor would make the subject unsuitable for inclusion, or could interfere with the subject participating in or completing the Study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2023-02-15 (Actual); Primary Completion 2024-07-29 (Actual); Study Completion 2024-07-29 (Actual)

PRIMARY OUTCOMES:
Incidence, severity and dose-relationship of AEs | 4 weeks
  Safety and tolerability of ARCT-032 assessed by determining the incidence, severity and dose-relationship of AEs by dose

SECONDARY OUTCOMES:
Change in plasma area under the curve after single dose of ARCT-032 | Up to 2 Weeks
  Area under the plasma concentration versus time curve (AUC) from time zero to the last quantifiable time point
Maximum observed plasma concentration (Cmax) after single dose of ARCT-032 | Up to 2 Weeks
  The maximum observed plasma concentration (Cmax)
Time at which Cmax occurred after single dose of ARCT-032 | Up to 2 Weeks
  The time at which Cmax occurred (Tmax)
AUC0-inf after single dose (Phase 1) or two doses (Phase 1b) of ARCT-032 | Up to 2 Weeks
  AUC from time zero extrapolated to infinity
T1/2 after single dose (Phase 1) or two doses (Phase 1b) of ARCT-032 | Up to 2 Weeks
  Terminal half-life
CL after single dose (Phase 1) or two doses (Phase 1b) of ARCT-032 | Up to 2 Weeks
  Total body clearance, calculated as dose divided by AUC0-inf
Vss after single dose (Phase 1) or two doses (Phase 1b) of ARCT-032 | Up to 2 Weeks
  Volume of distribution

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Program Director, Study Director — Arcturus Therapeutics
Locations (1):
- New Zealand Clinical Research, Christchurch, New Zealand

IPD SHARING:
Plan to Share IPD: No